CLINICAL TRIAL: NCT06244264
Title: A Single-center, Prospective, Randomized Controlled Study of the Safety and Efficacy of Autologous Transfusion in Spinal Surgery for Lung Cancer With Spinal Metastasis
Brief Title: The Safety and Efficacy of Autologous Transfusion in Spinal Surgery for Lung Cancer With Spinal Metastasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yu Zhang, PhD, Chief of Orthopedic Oncology, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPMAT001
Record Dates: First submitted 2024-01-15; First posted 2024-02-06 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Spinal Metastases; Blood Transfusion Complication; Lung Cancer; Surgery; Autologous Blood Transfusion
MeSH Terms: conditions — Transfusion Reaction; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: randomized parallel controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autoblood transfusion + leukocyte filter group (Experimental): In our department open surgery is considered as the standard procedure. The patients underwent open surgery, with autologous blood transfusion combined with a leukocyte filter. Blood transfusion based on bleeding during surgery.
  Interventions: Procedure: Autoblood transfusion
- Allogeneic blood transfusion group (No Intervention): In our department open surgery is considered as the standard procedure. The patients receives open surgery with allogeneic blood transfusion. Blood transfusion based on bleeding during surgery.

INTERVENTIONS:
Procedure: Autoblood transfusion — Through a negative pressure suction device, the patient's blood that flows out during surgery is collected into a blood storage filter. During the suction process, it is mixed with an appropriate anticoagulant and passed through multiple layers of filters. When the volume of recovered blood reaches a certain level, it is continuously (or intermittently) centrifuged. Using a high-speed centrifugal blood recovery tank, the red blood cells are separated, and the plasma, waste, cell fragments, anticoagulants, and harmful components are diverted into a waste bag. A large amount of saline is used to repeatedly wash, purify, and concentrate the red blood cells. Finally, the concentrated red blood cells are prepared into a 70% red blood cell suspension with saline and stored in a collection bag for transfusion back to the patients. Open surgery is considered as the standard procedure for metastatic spinal cord compression
  Arms: Autoblood transfusion + leukocyte filter group

SUMMARY:
The goal of this single-center prospective randomized controlled trial is to test and compare the safety and effectiveness of autologous blood transfusion in spinal surgery for lung cancer spinal metastases. The main questions it aims to answer are:

* Does autologous blood transfusion increase the incidence of new metastases?
* Does autologous blood transfusion affect postoperative hemoglobin levels and the number of circulating tumor cells in the blood?
* Can autologous blood transfusion reduce the rate of allogeneic transfusion during and after surgery for spinal metastases?

DETAILED DESCRIPTION:
In this study, participants underwent standard open spinal decompression surgery, and when blood transfusion was needed, autologous blood transfusion or allogeneic blood transfusion was used. Participants will be patients with lung cancer spinal metastases. Investigators will use flow cytometry, immunohistochemistry, and tumor cell culture methods to measure the number of circulating tumor cells in the blood before and after autologous blood transfusion.

Investigators will compare participants who receive autologous blood transfusion with those who do not to observe if there are differences in:

* The incidence of new metastases
* The rate of allogeneic transfusion during and after surgery
* Postoperative hemoglobin levels
* The number of circulating tumor cells in the blood
* The cost associated with transfusion

ELIGIBILITY:
Inclusion Criteria:

* The age range is 18-75 years old;
* The pathological diagnosis was lung cancer and spinal metastatic tumor;
* Expected survival > 3 months, can tolerate surgery;
* Unstable spine; And/or spinal cord nerve compression, nerve function; Progressive decline, palliative spinal open decompression surgery
* Patients with intraoperative/postoperative Hb<90 g/L or other conditions requiring blood transfusion

Exclusion Criteria:

* Serious heart dysfunction or heart failure, diagnosed blood system diseases, coagulation disorders;
* Severe renal insufficiency or need hemodialysis treatment;
* Sepsis or septicemia;
* Unable to obtain consent from the patient or family.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative and postoperative allogeneic blood transfusion rate | Through study completion, an average of 1 year
  The number of allogeneic blood transfusion patients (Intraoperative or postoperative )/ the total number of patients

SECONDARY OUTCOMES:
Number of circulating tumor cells in the blood | within 30 days post-surgery
  Number of circulating tumor cells in the blood
Incidence of transfusion related adverse reactions | within 14 days post-surgery
  the number of adverse reactions/ the total number of patients
occurence of new lesions | through study completion, an average of 1 year
  the number of patients with occurence of new lesions / the total number of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong provincial people's hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
After the research is completed, the data may be publicly shared depending on the outcome.